CLINICAL TRIAL: NCT06704724
Title: A PHASE 1 OPEN-LABEL STUDY OF PF-07985045 AS A SINGLE-AGENT AND IN COMBINATION WITH OTHER ANTI-CANCER AGENTS IN PARTICIPANTS WITH ADVANCED SOLID TUMORS
Brief Title: A Study to Learn About the Study Medicine PF-07985045 When Given Alone or With Other Anti-cancer Therapies in People With Advanced Solid Tumors That Have a Change in a Gene.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C6081001; 2024-517988-23-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Pancreatic Ductal; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Pancreatic Ductal; Carcinoma, Ductal, Pancreatic; Duct-Cell Carcinoma of the Pancreas; Duct-Cell Carcinoma, Pancreas; Ductal Carcinoma of the Pancreas; Pancreatic Duct Cell Carcinoma; Pancreatic Ductal Carcinoma; pancreatic ductal adenocarcinoma; PDAC; Colorectal Neoplasms; Colorectal Cancer; Colorectal Carcinoma; Colorectal Tumors; Neoplasms, Colorectal; Rectal Cancer; Colon Cancer; CRC; MSS CRC; Carcinoma, Non-Small-Cell Lung; Non-Small Cell Lung Cancer; Non-Small Cell Lung Carcinoma; Non-Small-Cell Lung Carcinoma; Nonsmall Cell Lung Cancer; Lung Cancer; NSCLC; KRAS; KRAS gene mutation
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Rectal Neoplasms; Colonic Neoplasms; Lung Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Cetuximab; Fluorouracil; Oxaliplatin; Leucovorin; Bevacizumab; pembrolizumab; Pemetrexed; Cisplatin; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Part 1 Dose Escalation (Experimental): PF-07985045 monotherapy Dose Escalation at prescribed dose and frequency in 28-day cycles
  Interventions: Drug: PF-07985045
- Part 1 Cohort A1 (Experimental): PF-07985045 monotherapy dose expansion in 2-3L PDAC at prescribed dose and frequency in 28-day cycles
  Interventions: Drug: PF-07985045
- Part 1 Cohort B1 (Experimental): PF-07985045 monotherapy dose expansion in 2-3L CRC at prescribed dose and frequency in 28-day cycles
  Interventions: Drug: PF-07985045
- Part 1 Cohort C1 (Experimental): PF-07985045 monotherapy dose expansion in 2-3L NSCLC at prescribed dose and frequency in 28-day cycles
  Interventions: Drug: PF-07985045
- Part 1 Cohort D1 (Experimental): PF-07985045 monotherapy dose expansion in other tumor types at prescribed dose and frequency in 28-day cycles
  Interventions: Drug: PF-07985045
- Part 2 Cohort A2 (Experimental): Combination (PF-07985045 + Gemcitabine + Nab-paclitaxel) dose escalation/expansion in 1L PDAC.
  Prescribed dose and frequency in 28-day cycles
  Interventions: Drug: PF-07985045; Combination Product: Gemcitabine; Combination Product: Nab-paclitaxel
- Part 2 Cohort B2 (Experimental): Combination (PF-07985045 + Cetuximab) dose escalation/expansion in 2-3L CRC
  Prescribed dose and frequency in 28-day cycles
  Interventions: Drug: PF-07985045; Combination Product: Cetuximab
- Part 2 Cohort B3 (Experimental): Combination (PF-07985045 + FOLFOX + Bevacizumab) dose escalation/ expansion in 1L CRC
  Prescribed dose and frequency in 28-day cycles
  Interventions: Drug: PF-07985045; Combination Product: Fluorouracil; Combination Product: Oxaliplatin; Combination Product: Leucovorin; Combination Product: Bevacizumab
- Part 2 Cohort B4 (Experimental): Combination (PF-07985045 + FOLFOX + Cetuximab) dose escalation/ expansion in 1L CRC
  Prescribed dose and frequency in 28-day cycles
  Interventions: Drug: PF-07985045; Combination Product: Cetuximab; Combination Product: Fluorouracil; Combination Product: Oxaliplatin; Combination Product: Leucovorin
- Part 2 Cohort C2 (Experimental): Combination (PF-07985045 + Pembro or sasanlimab) dose escalation/expansion in 1L NSCLC (TPS ≥ 50%)
  Prescribed dose and frequency in 21-day (pembro) or 28-day (sasanlimab) cycles
  Interventions: Drug: PF-07985045; Combination Product: Pembrolizumab; Combination Product: Sasanlimab
- Part 2 Cohort C3 (Experimental): Combination (PF-07985045 + Pembro + Platinum Chemo) dose escalation/expansion in 1L NSCLC (any TPS)
  Prescribed dose and frequency in 21-day cycles
  Interventions: Drug: PF-07985045; Combination Product: Pembrolizumab; Combination Product: pemetrexed; Combination Product: Cisplatin; Combination Product: Paclitaxel; Combination Product: Carboplatin
- Part 2 Cohort X (Experimental): Combination (PF-07985045 + PF-07284892) dose escalation/expansion
  Prescribed dose and frequency in 21-day cycles
  Interventions: Drug: PF-07985045; Combination Product: PF-07284892

INTERVENTIONS:
Drug: PF-07985045 — KRAS inhibitor
  Other Names: PF-5045
Combination Product: Gemcitabine — Chemotherapy (antimetabolite)
  Other Names: Gemzar
  Arms: Part 2 Cohort A2
Combination Product: Nab-paclitaxel — Taxane-type Chemotherapy
  Other Names: Abraxane
  Arms: Part 2 Cohort A2
Combination Product: Cetuximab — Monoclonal Antibody (EGFR Inhibitor)
  Other Names: Erbitux
  Arms: Part 2 Cohort B2; Part 2 Cohort B4
Combination Product: Fluorouracil — Part of FOLFOX chemotherapy regimen
  cytotoxic chemotherapy (antimetabolite and pyrimidine analog)
  Other Names: 5-FU; 5-fluorouracil
  Arms: Part 2 Cohort B3; Part 2 Cohort B4
Combination Product: Oxaliplatin — Part of FOLFOX Chemotherapy Regimen
  platinum based compound (alkylating agent)
  Other Names: Eloxatin
  Arms: Part 2 Cohort B3; Part 2 Cohort B4
Combination Product: Leucovorin — Part of FOLFOX chemotherapy regimen
  Folic Acid Analog
  Other Names: Folinic Acid; Wellcovorin; calcium folinate; Leucovorin Calcium
  Arms: Part 2 Cohort B3; Part 2 Cohort B4
Combination Product: Bevacizumab — VEG-F inhibitor
  Other Names: Zirabev; Avastin
  Arms: Part 2 Cohort B3
Combination Product: Pembrolizumab — immune checkpoint inhibitor (PD-1 inhibitor
  Other Names: Pembro; Lambrolizumab; MK-3475; Keytruda
  Arms: Part 2 Cohort C2; Part 2 Cohort C3
Combination Product: Sasanlimab — immune checkpoint inhibitor (PD-1 inhibitor)
  Other Names: PF-06801591
  Arms: Part 2 Cohort C2
Combination Product: pemetrexed — Can be used in Platinum-based Chemotherapy regimen
  Antimetabolite
  Other Names: Alimta
  Arms: Part 2 Cohort C3
Combination Product: Cisplatin — Can be used as part of Platinum-based chemotherapy regimen
  Platinum-based antineoplastic (alkylating agent)
  Other Names: Platinol; Cisplatinum; neoplatin
  Arms: Part 2 Cohort C3
Combination Product: Paclitaxel — Can be used in Platinum-based chemotherapy regimen
  Taxane
  Other Names: Taxol; Onxol
  Arms: Part 2 Cohort C3
Combination Product: Carboplatin — Can be used as part of a platinum-based chemotherapy regimen
  platinum containing compound (alkylating agent)
  Other Names: Paraplatin; Stricarb
  Arms: Part 2 Cohort C3
Combination Product: PF-07284892 — PF-07284892 used as a combination product.
  Other Names: ARRY-558
  Arms: Part 2 Cohort X

SUMMARY:
The purpose of this study is to learn about the safety and effects of the study medicine when given alone or together with other anti-cancer therapies. Anti-cancer therapy is a type of treatment to stop the growth of cancer.

This study also aims to find the best amount of study medication.

This study is seeking participants who have solid tumors (a mass of abnormal cells that forms a lump or growth in the body) that:

* are advanced (cancer that doesn't disappear or stay away with treatment) and
* have a KRAS gene mutation (a change in the DNA of the KRAS gene that can cause cells to grow in very high numbers).

This includes (but limited to) the following cancer types:

* Non-Small Cell Lung Cancer (NSCLC): It's a type of lung cancer where the cells grow slowly but often spread to other parts of the body.
* Colorectal Cancer (CRC): This is a disease where cells in the colon (a part of large intestine) or rectum grow out of control.
* Pancreatic ductal adenocarcinoma (PDAC): This is a cancer that starts in the ducts of the pancreas but can spread quickly to other parts of the body. Pancreas is a long, flat gland that lies in the abdomen behind the stomach. Pancreas creates enzymes that help with digestion. It also makes hormones that can help control your blood sugar levels.

All participants in this study will take the study medication (PF-07985045) as pill by mouth. This will be repeated for 21-day or 28-day cycles.

Depending on which part of the study participants are enrolled into they will receive the study medication (PF-07985045 alone or in combination with other anti-cancer medications). These anti-cancer medications will be given in the study clinic by intravenous (IV) that is directly injected into the veins at different times (depending on the treatment) during the 21-day or 28-day cycle.

Participants can continue to take the study medication (PF-07985045) and the combination anti-cancer therapy until their cancer is no longer responding.

The study will look at the experiences of people receiving the study medicines. This will help see if the study medicines are safe and effective.

Participants will be in this study for up to 4 years. During this time, the participants will come into the clinic for 1 to 4 times in each 21-day or 28-day cycle. After the participants have stopped taking the study medication (at about at 2 years) they will be followed for another two years to see how they are doing

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of advanced, unresectable, and/or metastatic or relapsed/refractory solid tumor.

  * Note for PDAC: Only participants with the histologic type of adenocarcinoma of the pancreas are allowed to enroll. For PDAC, if loco-regional disease is present, must also have metastatic disease.
  * Note for NSCLC: If a driver mutation is present, the participant was resistant or intolerant of precision medicine therapy (eg, inhibitors of EGFR, ALK, ROS1, or others).
* ECOG PS 0 or 1
* Presence of at least 1 measurable lesion based on RECIST version 1.1 that has not been previously irradiated.
* Documentation of mutated KRAS gene

  a. KRAS mutations of any variant except previously treated with any KRAS inhibitor
* Part 1: Participant must have progressed on standard treatment(s) for which no additional, effective therapy is available.

  1. PDAC (2-3L): Participants must have received and radiologically progressed on prior lines of systemic therapy for metastatic pancreatic adenocarcinoma. If participants received prior neoadjuvant or adjuvant chemotherapy and progressed within 6 months of the last dose, then this should be considered as a prior line of systemic therapy.
  2. NSCLC (2-3L): Participants must have received prior lines of anti-cancer treatment and progressed on at least a platinum-containing chemotherapy regimen and/or checkpoint inhibitor therapy; for participants with EGFR, ALK, or other genomic tumor alterations, participants must have progressed on approved therapy for these alterations.
  3. CRC (2-3L): Participants must have had only one or two prior systemic treatment regimens for mCRC. For either one or two prior treatments, these regimens must have included a fluoropyrimidine, oxaliplatin, or irinotecan; for one prior treatment, exposure to VEGF/VEGF receptor (VEGFR) inhibitor is optional.
  4. other tumors: Participants, in the judgment of the investigator, must have progressed or become intolerant to all available standard therapies, or have refused such therapy.
* Part 2:

  1. PDAC (1L) Cohort A2: Participants must not have received prior chemotherapy for metastatic disease. Participant could have received neoadjuvant therapy, adjuvant therapy, or adjuvant chemo-radiotherapy, as long as relapse did not occur within 6 months of completing these forms of adjuvant treatment. If so, the relapse within 6 months would be considered a line of therapy; the participant would be considered 2L, and not 1L.
  2. CRC (2-3L) Cohort B2: Participants must have had one or two prior systemic treatment regimens for mCRC. For either one or two prior treatments, these regimens must have included a fluoropyrimidine, irinotecan, oxaliplatin; for one prior treatment, exposure to a VEGF/VEGF receptor (VEGFR) inhibitor is optional.
  3. CRC (1L) Cohort B3: Participants must not have had prior chemotherapy for advanced or metastatic disease. Participant could have received adjuvant chemotherapy or adjuvant chemo-radiotherapy, as long as relapse did not occur within 6 months of complete of adjuvant therapy. If so, the relapse within 6 months would be considered a line of therapy; the participant would be considered 2L, and not 1L.
  4. NSCLC (1L) Cohort C2: Participants must have a TPS ≥50% and must not have received prior systemic treatment setting.
  5. NSCLC (1L) Cohort C3: Participants with any TPS and must not have received prior systemic treatment setting.

Exclusion Criteria:

* Active pneumonitis/ILD, pulmonary fibrosis requiring treatment with systemic steroid therapy. Additionally, participants in IO combinations (Cohorts C2 and C3) with history and/or active pneumonitis/ILD or pulmonary fibrosis requiring steroids are excluded from enrollment.
* Active or history of clinically significant gastrointestinal (GI) disease (including but not limited to inflammatory GI disease [eg, ulcerative colitis, Crohn's disease, inflammatory bowel disease], immune-mediated colitis, peptic ulcer disease, GI bleeding, chronic diarrhea) and other conditions that are unresolved and/or may increase the risk associated with study participation or study treatment administration.
* Active bleeding disorder, including GI bleeding, as evidenced by hematemesis, significant hemoptysis or melena in the past 6 months.
* Major surgery or completion of radiation therapy ≤4 weeks prior to enrollment/randomization or radiation therapy that included >30% of the bone marrow.
* Has symptomatic ascites or pleural effusion. A participant who is clinically stable following treatment for these conditions (including drainage catheter placement, therapeutic thoracentesis or abdominal paracentesis) is eligible.
* Current use or have received PPIs in the last seven days prior to starting study treatment.
* Known sensitivity or contraindication to any component of study intervention (PF-07985045, gemcitabine, nab-paclitaxel, cetuximab, bevacizumab, FOLFOX, 5-FU, pembrolizumab, sasanlimab, cisplatin, carboplatin, pemetrexed, SHP2 inhibitor(s).
* Hematologic abnormalities.
* Renal impairment.
* Hepatic abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2028-03-11 (Estimated); Study Completion 2029-03-11 (Estimated)

PRIMARY OUTCOMES:
Part 1 & 2: Incidence of Adverse Events (AEs) | Start of treatment up to 30 days after last dose or start of new anticancer therapy (whichever occurs first)
  An adverse event (AE) was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship to it. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/ incapacity; congenital anomaly. AEs included both serious and all non-serious AEs.
PART 1 & 2: Number of participants with laboratory abnormalities | From start of treatment up to 30 days after last dose or start of new anticancer therapy, whichever occurred first
  Number of participants with laboratory test abnormalities. Laboratory test parameters included hematology, coagulation, liver function, renal function, electrolytes, clinical chemistry, and urinalysis (dipstick and microscopy).
Part 1 & Part 2 (Dose Escalation Only): Number of participants with Dose-limiting toxicities (DLT) | Baseline up to 28 days
  Any of the prespecified AEs that are attributable to one, the other, or both study treatments, occurring in the DLT observation period are considered DLTs, excluding toxicities clearly due to underlying disease or extraneous causes
Part 2: Objective Response - Number of Participants With Objective Response (alone or in combination) | Baseline and every 8 to 12 weeks through time of confirmed disease progression, death, unacceptable toxicity, or through study completion, approximately 2 years'
  Percentage of participants with objective response-based assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) for overall response rate (ORR) assessed by the Investigator.

SECONDARY OUTCOMES:
Part 1 & 2: Maximum Observed Serum Concentration (Cmax) | baseline through end of Cycle 1 (All cycles are 28 days except Part 2 Cohort C2/C3 which are 21 days)
  Evaluate the single and multiple dose PK ofPF-07985045 as monotherapy, or in combination with other anti-tumor agents.
Part 1& 2: Time to Reach Maximum Observed Serum Concentration (Tmax) | Baseline through end of Cycle 1 (All cycles are 28 days except part 2 Cohort C2/C3 which are 21 days)
  Evaluate the single and multiple dose PK of PF-07985045 as monotherapy, or in combination with other anti-tumor agents.
Part 1 & 2: Serum Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | Baseline through end of Cycle 1 (All cycles are 28 days except Part 2 Cohort C2/C3 which are 21 days)
  Evaluate the single and multiple dose PK of PF-07985045 as monotherapy, or in combination with other anti-tumor agents.
Part 1 & 2: Changes in pERK levels | Baseline through end of Cycle 1 (All cycles are 28 days except Part 2 Cohort C2/C3 which are 21 days)
  Evaluates the intended mechanism of action (MoA) modulation of KRAS inhibition and target engagement effect of PF-07985045 in peripheral blood of participants with advanced solid tumor malignancies.
Objective Response - Number of Participants With Objective Response | Baseline and every 8 to 12 weeks through time of confirmed disease progression, death, unacceptable toxicity, or through study completion, approximately 2 years
  Percentage of participants with objective response-based assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) assessed by the Investigator including overall response rate (ORR) (Part 1 only), progression free survival (PFS), and duration of response (DOR).
Part 1: Effect of Food on Cmax | Baseline through end of Cycle 1 (All cycles are 28 days)
  Evaluate the effect of food on Cmax of PF-07985045 as monotherapy.
Part 1: Effect of Food on Tmax | Baseline through end of Cycle 1 (All cycles are 28 days)
  Evaluate the effect of food on Tmax of PF-07985045 as monotherapy.
Part 1: Effect of Food on AUClast | Baseline through end of Cycle 1 (All cycles are 28 days)
  Evaluate the effect of food on AUClast of PF-07985045 as monotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (15):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - City of Hope (City of Hope National Medical Center, City Of Hope Medical Center), Duarte, California
  - City of Hope Investigational Drug Service (IDS), Duarte, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - DFCI Chestnut Hill, Newton, Massachusetts
  - Columbia University Irving Medical Center, New York, New York
  - CUMC Research Pharmacy, New York, New York
  - The Trustees of Columbia University and The New York and Presbyterian Hospital, New York, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Board of Regents of the University of Wisconsin System, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center-University Hospital, Madison, Wisconsin
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Shizuoka Cancer Center, Nagaizumi-cho, Shizuoka
- Pan American Center for Oncology Trials, LLC, Rio Piedras, Puerto Rico

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C6081001